CLINICAL TRIAL: NCT04166682
Title: A Study of the Impact of Home-based Cardiac Rehabilitation on Outcomes After Transcatheter Aortic Valve Replacement (TAVR)
Brief Title: Impact of Home-based Cardiac Rehabilitation on Outcomes After TAVR
Acronym: HBCR-TAVR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ZJUWXY
Record Dates: First submitted 2019-08-26; First posted 2019-11-18 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2019-07

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Routine care
  Interventions: Behavioral: Routine care
- Interventional Group (Experimental): Home-based cardiac rehabilitation
  Interventions: Behavioral: Home-based cardiac rehabilitation

INTERVENTIONS:
Behavioral: Home-based cardiac rehabilitation — cardiac rehabilitation done at home
  Arms: Interventional Group
Behavioral: Routine care — Routine care and followup
  Arms: Control Group

SUMMARY:
To evaluate the effects of a home-based cardiac rehabilitation program for Chinese patients after Transcatheter Aortic Valve Replacement (TAVR).

ELIGIBILITY:
Inclusion Criteria:

* Aortic stenosis accepted for TAVR
* Participant able and willing to give written informed consent
* Participant able (in the investigator's opinion) and willing to comply with all study requirements

Exclusion Criteria: subjects may not enter the study if any of the following apply

* Intervention deemed inappropriate due to co-morbidity or frailty
* Life expectancy less than one year due to co-morbidity
* Previous surgical aortic valve replacement (sAVR) or TAVR
* Predominant aortic regurgitation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-05-09 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test | 6 weeks
  The total distance walked in meters during 6 minutes.

SECONDARY OUTCOMES:
Number of participants die | 6 weeks, 12 months
  Number of participants die during the study due to cardiovascular or non-cardiovascular causes.
Number of participants rehospitalized | 6 weeks, 12 months
  Number of participants rehospitalized during the study.
Number of participants completing home-based cardiac rehabilitation | 6 weeks
  Number of participants completing home-based cardiac rehabilitation
Cardiac function | 12 months
  Ejection fraction estimated by echocardiography
Aortic valve function | 12 months
  Aortic valve function estimated by echocardiography
Number of participants injured | 6 weeks
  Number of participants injured or die during the course of home-based cardiac rehabilitation
Time spent performing activities | 6 weeks, 12 months
  Number of minutes in a typical week that participants spent performing activities
6-minute walk test | 12 months
  The total distance walked in meters during 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Xianbao Liu, Doctor, Study Chair — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- The second affiliated hospital of zhejiang university, school of medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abraham LN, Sibilitz KL, Berg SK, Tang LH, Risom SS, Lindschou J, Taylor RS, Borregaard B, Zwisler AD. Exercise-based cardiac rehabilitation for adults after heart valve surgery. Cochrane Database Syst Rev. 2021 May 7;5(5):CD010876. doi: 10.1002/14651858.CD010876.pub3. PMID 33962483